CLINICAL TRIAL: NCT06291961
Title: A Single-arm, Open-label Phase I Clinical Trial to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamic Profile of a Single Dose of CS-101 Injection in Subjects With β-thalassemia Major
Brief Title: A Safety and Efficacy Study Evaluating CS-101 in Subjects With β-Thalassemia Major
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CorrectSequence Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-101-01
Record Dates: First submitted 2024-02-23; First posted 2024-03-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Beta-Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS-101 injection (Experimental): Autologous CD34+ hematopoietic stem cell suspension modified by in vitro base editing technique
  Interventions: Genetic: CS-101 injection

INTERVENTIONS:
Genetic: CS-101 injection — Autologous CD34+ hematopoietic stem cell suspension modified by in vitro base editing technique

SUMMARY:
The goal of this open label, single-arm clinical study is to learn about the safety and efficacy of CS-101 in treating patients with β-thalassemia major anemia.

DETAILED DESCRIPTION:
CS-101 is an autologous CD34+(Cluster of differentiation 34) cell suspension, edited by in vitro base editing technology, which modifies the BCL11A(B-cell lymphoma/leukemia 11A) binding site in HBG(Hemoglobin Subunit Gamma) promoter, so that it loses the ability to bind to BCL11A, which can re-induce the production of γ-globin chain and increase the concentration of HbF(fetal hemoglobin) in the blood, compensating for the function of missing HbA(adult hemoglobin) to achieve clinical cure. The therapy addresses two major challenges in the current treatment of the disease: lack of matching donors and graft-versus-host diseases in allogeneic hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 35 years old(inclusive) male or female subjects at the time of informed consenting. For minors, their legal representative is required to sign the informed consent form, besides, if the subjects aged 8 years or older, they should provide a signed and dated.
* Diagnosis of β-thalassemia major.
* Generally in good condition, Karnofsky performance score≥60 points for subjects≥16 years old, or Lansky Play-Performance score≥60 points for subjects under 16 years old.
* For female subjects of childbearing potential: use effective contraceptive measures from the start of screening and agree to continue using such measures for contraception throughout the study
* For male subjects who have a potential ability to father a child: use condoms or other methods continuously from the start of mobilization to ensure effective contraception for sexual partners during the study period

Exclusion Criteria:

* Treatment with other investigational medications or other experimental interventions 30 days prior to signing informed consent or within 6 half-lives of the drug, whichever is longer
* Subjects who have received or are receiving thalidomide and/or Luspatercept in the past 6 months before screening
* Previously received allogeneic hematopoietic stem cell transplantation or gene(edited) therapy
* Subjects have available related fully matching donors and are eligible and prepared for allogeneic hematopoietic stem cell transplantation
* Patients with coexisting α-thalassemia and more than 2 deletions or non-deletional mutations in the α-globin chain coding genes
* Known to be allergic to drugs used during autologous hematopoietic stem cell transplantation (including but not limited to granulocyte colony-stimulating factor, busulfan, dextran), excipients(such as dimethyl sulfoxide), or instruments(such as intravenous catheters) as determined by the investigator are deemed unsuitable to participate in this study
* Those with positive results in HIV, cytomegalovirus, Epstein-Barr virus and treponema pallidum test, active infection of hepatitis B, hepatitis C, or known tuberculosis, parasitic infection, etc. Hepatitis B stabilized on medication(HBV-DNA test negative) and cured hepatitis C(HCV-RNA test negative) can be considered acceptable.
* Echocardiography shows ejection fraction below 45%
* Laboratory indicators, defined as：Aspartate aminotransferase(AST), alanine aminotransferase(ALT) >3× upper limit of normal(ULN) or Baseline International Normalized Ratio(INR)>1.5×ULN.
* MRI during the screening period shows severe cardiac iron overload and other conditions, and are judged by the investigator to be intolerable or inappropriate for autologous hematopoietic stem cell transplantation
* Patients with past/present history of cancer
* Known neurological disorders, psychological problems or mental illness, and is judged by the investigator to be unable to cooperate with the study procedures
* Known history of uncontrolled epileptic seizures and is judged by the investigator to be unfit to participate in this study
* The investigators determined that a non-hypersplenism-induced white blood cell count of<3×10^9/L, and/or a platelet count of<100×10^9/L.
* Known history of other serious cardiovascular, pulmonary, renal diseases, digestive tract conditions, liver diseases and / or other conditions, etc., and are judged by the investigator to be intolerable or inappropriate for autologous hematopoietic stem cell mobilization, collection, and myeloablative conditioning and infusion
* Pregnant or lactating women

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
AEs(Adverse Events) and SAEs(Serious Adverse Events) after CS-101 infusion | From signing informed consent to 12 months post-CS-101 infusion
  Frequency and severity of adverse events(AEs）as assessed by CTCAE(Common Terminology Criteria for Adverse Events)v5.0
Overall survival rate | Up to 12 months post-CS-101 infusion
Proportion of subjects with engraftment | Within 42 days post-CS-101 infusion
  Subjects with engraftment is defined as neutrophil engrafted
Time to neutrophil engraftment | Up to 12 months post-CS-101 infusion
  Time to neutrophil engraftment is defined as first day of 3 consecutive measurements of absolute neutrophil count≥0.5×10^9/L on three different days.
Time to platelet engraftment | Up to 12 months post-CS-101 infusion
  Time to platelet engraftment is defined as first day of 3 consecutive measurements of absolute platelet count≥20×10^9/L on three different days and without platelet transfusion.
Incidence of transplant-related mortality | From baseline to 100 days post-CS-101 infusion
  Incidence of transplant-related mortality(Transplant-related mortality events defined as deaths assessed by the investigator as potentially transplant-related)
Change in fetal hemoglobin(HbF) concentration over time | Up to 12 months post-CS-101 infusion
  Fetal hemoglobin(HbF) concentration from baseline to 9 months post-CS-101 infusion
Change in total hemoglobin(Hb) concentration over time | Up to 12 months post-CS-101 infusion
  Total hemoglobin concentration change from baseline to 9 months post-CS-101 infusion

SECONDARY OUTCOMES:
Chimerism level in Peripheral blood and bone marrow | Up to 12 months post-CS-101 infusion
  Proportion of alleles with intended genetic modification in peripheral blood leukocytes and bone marrow over time
Proportion of subjects achieving transfusion independence for at least 6 consecutive months | From CS-101 infusion up to 12 months post-CS-101 infusion
  Maintaining transfusion independence for at least 6 consecutive months while maintaining a weighted mean hemoglobin≥9 g/dL Proportion of subjects
Proportion of subjects achieving fetal hemoglobin(HbF) increase≥2.0 g/dL | Up to 2 months post-CS-101 infusion
  Fetal hemoglobin(HbF) concentration increase≥2.0 g/dL within 2 months post-CS-101 infusion
Proportion of subjects achieving fetal hemoglobin(HbF) increase≥7.0 g/dL | Up to 6 months post-CS-101 infusion
  Fetal hemoglobin(HbF) concentration increase≥7.0 g/dL within 6 months post-CS-101 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Yaliang Li, Study Director — CorrectSequence Therapeutics Co., Ltd
Locations (3):
- China (3):
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Ruijin Hospital Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality